CLINICAL TRIAL: NCT03449810
Title: Effectiveness of Muscles Energy Technique on Quality of Life and Trunk Muscles Functions in Patients With Chronic Non-specific Low Back Pain
Brief Title: Effectiveness of Muscles Energy Technique in the Management of Chronic Non-specific Low Back Pain
Acronym: MET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of KwaZulu (Other)
Responsible Party: Principal Investigator, Usman Ahmed, Principal Investigator, University of KwaZulu
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 217077488
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Chronic Non-specific Low Back Pain
Keywords: MET, Low Back Pain, Stabilization exercises; Quality of Life, Functional disability
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: The Intervention Models Includes; Muscles Energy Technique plus Dynamic stabilization exercises which would be administered to participants in group A, Dynamic stabilization exercises to be administered to group B participants and group C which is the control will receive standard physiotherapy treatment.
Who Masked: Participant, Outcomes Assessor
Masking Description: All eligible participants will be randomly be allocated to three groups using a random number generator by an independent person (third party). Two study assessors will take measurements of all outcomes at baseline, 6th and 12th week and 3 months follow-up, however, they will be blinded to group allocation. Group indication will be placed in a sealed envelope that will be opened after the study assessors have performed the initial assessments and the participants will be instructed not to disclose their study groups to the assessors. However, participants are expected to be unaware of their group procedure/intervention, therefore, the physiotherapists will be instructed not to disclose the name of their group procedure to the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DSE plus MET (group A) (Experimental): The DSE will consist of seven exercise activities that will be administered at random viz; 1. Bridging 2. Supine twist stretch 3. Double leg knee to chest stretch 4. Plank heel raise 5. Ball squat 6. Leg press on ball 7. Hip Lifts.
  The MET procedure will involve a total of 5-10 contralateral isometric voluntary contractions that will be resisted by force equal to the participant's for 30 seconds with 5 seconds rest between contractions (corresponding to 20-30%).
  Interventions: Procedure: DSE plus MET group A
- DSE only (group B) (Active Comparator): The DSE will consist of seven exercise activities that will be administered at random viz; 1. Bridging 2. Supine twist stretch 3. Double leg knee to chest stretch 4. Plank heel raise 5. Ball squat 6. Leg press on ball 7. Hip Lifts.
  Interventions: Procedure: DSE alone group B
- Standard Physiotherapy Treatment (group C) (Active Comparator): This group will involve classical massage, therapeutic exercises (strengthening spinal and abdominal muscles) and a combination of interferential therapy and therapeutic ultrasound (INF/UTS) applied to the lumbosacral region. The participants will be asked to perform the therapeutic exercises once a day at home.
  Interventions: Procedure: Standard Physiotherapy treatment group C

INTERVENTIONS:
Procedure: DSE plus MET group A — The Dynamic stabilization exercises will consist of seven exercises, which are aimed to strengthen the lumbar stabilizing muscles. All seven dynamic stabilization exercises will be performed once and always in random order.
  The procedure for MET involves voluntary contraction of the participant's muscle in a precisely controlled direction, at varying levels of intensity, against a distinctly executed counterforce applied by the therapist. In this type of therapy, a participant contracts muscles by pushing against resistance provided by the therapist. The therapist then assists the participant in stretching, strengthening and relaxing those muscles.
  Arms: DSE plus MET (group A)
Procedure: DSE alone group B — The DSE in this arm is the same a described in group A, i.e. it involves seven exercises activities administered randomly at every session of the study intervention.
  Arms: DSE only (group B)
Procedure: Standard Physiotherapy treatment group C — In the control group, the participants will receive standard physiotherapy treatment offered for the management of chronic NSLBP patients in Nigeria. Therefore, individuals randomized to this therapeutic group will be treated with classical massage, therapeutic exercises and a combination of interferential therapy and therapeutic ultrasound (INF/UTS) applied to the lumbosacral region.
  Arms: Standard Physiotherapy Treatment (group C)

SUMMARY:
Low back pain is the most common health problem that affects work performance and quality of life. Non-specific low back pain (NSLBP) is defined as low back pain not attributable to a recognizable, known specific pathology. NSLBP is the leading cause of disability among the major musculoskeletal conditions which leads to Impairments, Activity Limitations and participation restrictions. Therefore it becomes a psychosocial/economic burden on individuals, families, communities, industries and government. Existing literature shows globally 40% to 50% of people have LBP at some point in their lives and there exists a challenge in Africa on the best rehabilitation methods for low back pain management which could prevent chronic pain and disability. Therefore, this study aims to determine the effectiveness of MET when combined with DSE in the management of chronic NSLBP patients and to analyze the additional effect the MET procedure will provide relative to DSE.

DETAILED DESCRIPTION:
Low back pain (LBP) is arguably the most prevalent musculoskeletal condition found among both developed and developing nations. Broadly defined as pain or discomfort in the lumbar region of the spine it is the leading cause of activity limitations, resulting in significant losses in productivity at work and incurs billions of dollars in medical expenditure annually. The prevalence of LBP worldwide is estimated to be between 30 and 80% among the general population and has been found to increase with age. In addition, a higher prevalence of LBP has been associated with lower socioeconomic status and lower education levels. According to the Global Burden of Disease (GBD) 2010 study, LBP is currently the 6th highest burden on a list of 291 conditions and is the cause of more years lived with disability globally than any other disease. Affecting just about anyone, of any gender, race or socioeconomic background, LBP has a substantial impact on the overall and financial well-being of an individual and society.

Therefore, it was postulated that the burden of LBP would be greater in lower and middle-income countries like those situated in Africa. A recent systematic review and meta-analysis published in 2018 revealed that the lifetime, annual and point prevalence of LBP among African nations, was higher than the global LBP prevalence. The majority of the studies included in this meta-analysis were conducted in Nigeria, which is a lower-middle-income country. In Nigeria, the annual prevalence rate of LBP has been reported between 33% and 74%, mostly affecting workers. The prognosis after an acute episode of LBP is less favourable than once thought, as 60-80% of the patients will experience recurrence or persistence of this disabling condition.12 Despite the high incidence and prevalence of LBP, little is known about the precise causes. As a clear pathoanatomic diagnosis cannot be identified in 85% of the patients,13 LBP in these patients is labelled as non-specific (NSLBP).

Despite extensive research, the issue of spinal pain management still constitutes a challenge for physicians, physiotherapists, and researchers. There are many therapies claimed to be useful for the treatment of NSLBP, but most of these treatments have not been well investigated or have been found to have modest effects in terms of pain relief and improving disability. Conservative treatment remains the best choice and usually involves physiotherapy. Exercise therapy is one of the most used treatment strategies as it has shown to be effective in decreasing pain and disability, and can even induce functional changes of the back muscles. Although, exercise therapy in highly recommend by experts in treatment guidelines, the evidenced treatment effects remain low to moderate. It is, therefore, useful to further explore the effectiveness of treatments that may assist people with NSLBP. Another, non-invasive, safe and inexpensive treatment technique used by physiotherapists, osteopaths, chiropractors and manual therapists in the treatment of NSLBP is Muscle Energy Technique (MET). MET involves alternating periods of resisted muscle contractions and assisted stretching. Although it has been suggested that MET can be used to lengthen a shortened muscle, mobilize an articulation with restricted mobility, strengthen a physiologically weakened muscle and reduce localized oedema and passive congestion, the physiological mechanisms underlying the therapeutic effects of MET are currently unclear. Mechanisms of altered proprioception, motor programming and control have been proposed, but research is required to confirm these hypotheses. While MET is often used for the treatment of NSLBP, a recent Cochrane review concluded that there is lack of empirical evidence on its effectiveness in the management of chronic NSLBP. These conclusions were made not because of the lack of treatment effectiveness, but because the currently available studies have been generally performed in too small study samples and have a high risk of bias, producing unreliable answers about this therapy. In conclusion, the Cochrane review emphasized the need for larger, high-quality studies to determine the effectiveness and safety of MET in chronic NSLBP.

Therefore, the aims of this study are to determine the effectiveness of MET when combined with DSE in the management of chronic NSLBP patients and to analyze the additional effect the MET procedure will provide relative to DSE. Thus, the efficacy of the combination of MET plus DSE will be compared with outcomes of treatment with DSE or standard physiotherapy (SP) in the management of chronic NSLBP. The study will evaluate the effect of each intervention on trunk Range of Motion (ROM), muscle functions (limited to muscles strength, endurance, force and Maximal voluntary contraction [MVC]), Quality of Life (QoL), functional disability, activity limitations and participation restrictions.

The primary goal of this study is to evaluate the effects of MET in combination with DSE on quality of life and trunk muscles functions in patients with chronic NSLBP, however, the study involves the following as general goal that needs to be realized;

1. To conduct a systematic review (scoping) of the literature on the effectiveness of MET in the management NSLBP.
2. To cross-culturally adapt and psychometrically validate the Nigerian Hausa Version of Örebro Musculoskeletal Pain Screening Questionnaire.
3. To conduct an online survey to determine the knowledge and skills of Nigerian physiotherapist on the application of MET in the management of NSLBP.
4. To evaluate the working mechanism of MET on the trunk muscle function by studying several muscular properties (recruitment, endurance, fatigability, flexibility) in chronic NSLBP.
5. To conduct a randomized control trial (RCT) to determine the short-term (6 weeks, 12 weeks) and long term (3 months) effectiveness of MET in combination with DSE on back muscles function and on clinical outcomes of functionality (such as disability, quality of life, and activity and participation restrictions) in patients with chronic NSLBP.

Therefore, the RCT component of this research has the following objectives.

1. To determine the effectiveness of MET in combination with DSE in the management of chronic NSLBP patients by assessing their influencing on trunk muscles functions limited to trunk muscles endurance, Transverses abdominus muscles contraction rate, trunk ROM, QoL, functional disability, global rating of change scale (GROCS), activity limitations and participation restrictions.
2. To evaluate the additional effect of MET relative to DSE on the study outcomes in the management of chronic NSLBP patients.
3. To compare the therapeutic effect of MET plus DSE with outcomes of treatment with DSE or standard physiotherapy (SP) in the management of chronic NSLBP
4. To assess all outcomes at baseline, 6th week and 12th week of the study interventions.
5. To also conduct a 3 months follow-up evaluation on outcomes to determine if the intervention effect is retained within the period. The ultimate goal is to provide recommendations (based on the study findings) for the implementation and use of MET in the Nigerian Health Care System for the management of chronic NSLBP.

ELIGIBILITY:
Inclusion Criteria:

1. NSLBP history of about or more than 3 months and associated with referred lower extremity pain; pain in the lumbopelvic region;
2. Lumbar hypomobility; mobility deficits of the thorax and hip regions;
3. LBP not of specific origin diagnosed by a physician (due to fracture, tumours, malignancy, ankyloses, infections, and pregnancy);
4. Diminished trunk or pelvic region muscle strength and endurance;
5. Movement coordination impairments while performing community/work-related recreational or occupational activities.
6. Attending Outpatient clinics and Physiotherapy departments of Rasheed Shekoni Teaching Hospital Dutse and Federal medical centre Birnin-Kudu in Jigawa state, Northwest Nigeria.

Exclusion Criteria:

1. Chronic NSLBP with radiating pain due to nerve root involvement in physical examination.
2. Patients using immunosuppression or steroid medication.
3. Patients with persistent severe pain.
4. Patients with spinal deformities.
5. Patients with widespread neurological symptoms; patients with peritonitis as at the time of recruitment; patients with a history of lumbar surgery; patients diagnosed with carcinoma or organ disease; and patients with a history of severe rheumatic, orthopaedic, cardiovascular, systemic, metabolic or neurologic disorders.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-10-14 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Medical Outcomes Survey Short-Form-36 (SF-36) | 6 month
  Quality of Life (QoL) will be assessed with SF-36, The questionnaire is divided into 10 segments with a total of 36 questions. The segments involve Demography, General Health, Limitation of Activities, Physical Health Problem, Emotional Health Problem, Social Activities, Pain, Energy and Emotion, Social Activities and General Health.
Activity Limitation and Participation Restriction | 6 month
  Level of activity Limitation and Participation Restriction would be measured using Orebro Musculoskeletal Pain Screening Questionnaire.

SECONDARY OUTCOMES:
Basal Mass Index (Demographic data) | Once
  Using formula; Body weight/Height square.
Skin fold thickness for percentage body fat (Demographic data) | Once
  Skin fold calliper would be used to measure participants skin fold thickness
Transverse abdominus muscles contraction rate | 6 months
  Pressure biofeedback unit
Level of pain perception | 6 months
  Level of Pain Perception would be measured using pain numeric rating scale, it has a scale of 0-10-mm (0 means no Pain, 1-3 means mild pain, 4-7 means moderate pain and 8-10 means severe pain) and the minimally important change for the visual analog scale is 2 (using a 0-10 self-report scale). The patient is asked to make three pain ratings, corresponding to current, best and worst pain experienced over the past 24 hours. The average of the 3 scores will represent patient's level of pain perception.
Functional Disability | 6 months
  Level of Functional Disabilities of Participant resulting from CMLBP would be measured using Oswestry disability Index
Spine range of motion | 6 months
  Inclinometer would be used to measure trunk range of motion
Trunk extension endurance test | 6 months
  Biering-sorensen test
Trunk flexion endurance test | 6 months
  McGill's torso battery test
Trunk side flexion endurance test | 6 months
  McGill's torso battery test
Global Rating of Change Scale (GROC) | 6 months
  This scale will be used to evaluate the satisfaction of the participant with the study intervention in term of improvement on symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: USMAN ABBA AHMED, MASTERS, Principal Investigator — University of KwaZulu; Maharaj S Sonill, PhD, Study Chair — University of KwaZulu; Nadasan N Thaya, PhD, Study Director — University of KwaZulu
Locations (1):
- Rasheed Shekoni Specialist Hospital, Dutse, Jigawa State, Nigeria

IPD SHARING:
Plan to Share IPD: Undecided
We have not yet decided whether to share IPD, but we will when we find it convenient

REFERENCES:
- [Background] Koes BW, van Tulder MW, Thomas S. Diagnosis and treatment of low back pain. BMJ. 2006 Jun 17;332(7555):1430-4. doi: 10.1136/bmj.332.7555.1430. No abstract available. PMID 16777886
- [Background] Manusov EG. Evaluation and diagnosis of low back pain. Prim Care. 2012 Sep;39(3):471-9. doi: 10.1016/j.pop.2012.06.003. PMID 22958556
- [Background] Balague F, Mannion AF, Pellise F, Cedraschi C. Non-specific low back pain. Lancet. 2012 Feb 4;379(9814):482-91. doi: 10.1016/S0140-6736(11)60610-7. Epub 2011 Oct 6. PMID 21982256
- [Background] Hoy D, Bain C, Williams G, March L, Brooks P, Blyth F, Woolf A, Vos T, Buchbinder R. A systematic review of the global prevalence of low back pain. Arthritis Rheum. 2012 Jun;64(6):2028-37. doi: 10.1002/art.34347. Epub 2012 Jan 9. PMID 22231424
- [Background] Louw QA, Morris LD, Grimmer-Somers K. The prevalence of low back pain in Africa: a systematic review. BMC Musculoskelet Disord. 2007 Nov 1;8:105. doi: 10.1186/1471-2474-8-105. PMID 17976240
- [Background] Omokhodion FO. Low back pain in an urban population in Southwest Nigeria. Trop Doct. 2004 Jan;34(1):17-20. doi: 10.1177/004947550403400107. PMID 14959964
- [Background] Sikiru L, Shmaila H. Prevalence and risk factors of low back pain among nurses in Africa: Nigerian and Ethiopian specialized hospitals survey study. East Afr J Public Health. 2009 Apr;6(1):22-5. doi: 10.4314/eajph.v6i1.45737. PMID 20000059
- [Background] Cohen SP, Argoff CE, Carragee EJ. Management of low back pain. BMJ. 2008 Dec 22;337:a2718. doi: 10.1136/bmj.a2718. No abstract available. PMID 19103627
- [Background] Martell BA, O'Connor PG, Kerns RD, Becker WC, Morales KH, Kosten TR, Fiellin DA. Systematic review: opioid treatment for chronic back pain: prevalence, efficacy, and association with addiction. Ann Intern Med. 2007 Jan 16;146(2):116-27. doi: 10.7326/0003-4819-146-2-200701160-00006. PMID 17227935
- [Background] Mitchell, F. L., & Mitchell, P. K. G. (1999). The muscle energy manual, 4196(517), 48826.
- [Background] Franke H, Fryer G, Ostelo RW, Kamper SJ. Muscle energy technique for non-specific low-back pain. Cochrane Database Syst Rev. 2015 Feb 27;2015(2):CD009852. doi: 10.1002/14651858.CD009852.pub2. PMID 25723574
- [Background] Marshall PW, Murphy BA. Core stability exercises on and off a Swiss ball. Arch Phys Med Rehabil. 2005 Feb;86(2):242-9. doi: 10.1016/j.apmr.2004.05.004. PMID 15706550
- [Background] Hodges PW. Core stability exercise in chronic low back pain. Orthop Clin North Am. 2003 Apr;34(2):245-54. doi: 10.1016/s0030-5898(03)00003-8. PMID 12914264
- [Background] Charan J, Biswas T. How to calculate sample size for different study designs in medical research? Indian J Psychol Med. 2013 Apr;35(2):121-6. doi: 10.4103/0253-7176.116232. PMID 24049221
- [Background] Delitto A, George SZ, Van Dillen L, Whitman JM, Sowa G, Shekelle P, Denninger TR, Godges JJ; Orthopaedic Section of the American Physical Therapy Association. Low back pain. J Orthop Sports Phys Ther. 2012 Apr;42(4):A1-57. doi: 10.2519/jospt.2012.42.4.A1. Epub 2012 Mar 30. PMID 22466247
- [Background] Selkow NM, Grindstaff TL, Cross KM, Pugh K, Hertel J, Saliba S. Short-term effect of muscle energy technique on pain in individuals with non-specific lumbopelvic pain: a pilot study. J Man Manip Ther. 2009;17(1):E14-8. doi: 10.1179/jmt.2009.17.1.14E. PMID 20046557
- [Derived] Ahmed UA, Maharaj SS, Van Oosterwijck J. Effects of dynamic stabilization exercises and muscle energy technique on selected biopsychosocial outcomes for patients with chronic non-specific low back pain: a double-blind randomized controlled trial. Scand J Pain. 2021 Feb 24;21(3):495-511. doi: 10.1515/sjpain-2020-0133. Print 2021 Jul 27. PMID 33641272
- See also: Koes, B. W., Van Tulder, M. W., & Thomas, S. (2006). Diagnosis and Treatment of Low Back Pain. — http://doi.org/10.1136/bmj.332.7555.1430
- See also: Balagué, F., Mannion, A. F., Pellisé, F., & Cedraschi, C. (2012). Non-specific low back pain. — http://doi.org/10.1016/S0140-6736(11)60610-7
- See also: Louw QA, Morris LD, Grimmer-Somers K. The prevalence of low back pain in Africa: a systematic review — http://doi.org/10.1186/1471-2474-8-105
- See also: Sikiru, L., & Shmaila, H. (2009). Prevalence and risk factors of low back pain among nurses in Africa: Nigerian and Ethiopian specialized hospitals survey study — http://www.ncbi.nlm.nih.gov/pubmed/20000059
- See also: Cohen SP, Argoff CE, Carragee EJ. Management of low back pain. — http://doi.org/10.1136/bmj.a2718
- See also: Marshall, P. W., & Murphy, B. A. (2005). Core stability exercises on and off a Swiss ball. — http://doi.org/10.1016/j.apmr.2004.05.004
- See also: Hodges, P. W. (2003). Core stability exercise in chronic low back pain. — http://doi.org/10.1016/S0030-5898(03)00003-8
- See also: ANOVA power analysis — http://www.math.yorku.ca/SCS/Online/power/

DOCUMENTS (1):
  • Informed Consent Form (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/10/NCT03449810/ICF_000.pdf